CLINICAL TRIAL: NCT04668040
Title: Comparing the Effects of Stretching and Muscle Energy Technique in the Management of Lower Cross Syndrome
Brief Title: Comparison of Stretching and MET in Lower Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00383 Nouman Khan
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Cross Syndrome
Keywords: Muscle energy technique; Lower cross syndrome; stretching
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle energy technique (Experimental): Muscle energy technique applied in the lower cross syndrome muscle pattern.
  Interventions: Other: Muscle energy technique
- Stretching (Active Comparator): Stretching technique applied in the lower cross syndrome muscle pattern.
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Muscle energy technique — Muscle energy technique for illiopsoas, rectus femoris, erector spinae & hamstrings muscles duration of contraction was 10 sec, rest interval was 5 sec, stretch duration was 30 sec, number of repetition of stretch was 5, number of set was 1, frequency per week was 3
  Arms: Muscle energy technique
Other: Stretching — Stretching exercises for illiopsoas, rectus femoris, erector spinae & hamstrings muscles duration of stretch was 15 sec, rest interval was 5 sec, number of repetition was 5, number of set was 1, frequency per week was 3
  Arms: Stretching

SUMMARY:
The aim of the study is to compare the effects of stretching exercises & muscle energy techniques in the management of lower cross syndrome and to find the effective treatment in the lower cross syndrome management.

DETAILED DESCRIPTION:
In 2015 the systematic review estimated that prevalence of Chronic low back pain in 24 to 39 year old individual was 4.2% and the individual between 20 to 59 was 19.6% . The genesis and perpetuation of Low back pain (LBP) has many underlying factors among which one is proposed by Janda's concept of pelvic crossed syndrome. This condition describes a pattern of tight and weak muscles around the pelvis. Marked postural deviation is seen such as increased lumber lordosis and depending on this lordosis the muscle involvement can be distinguished. The center of the gravity is slightly anterior to S1 or S2, which means pelvis position, is key to faulty or good alignment.

Various studies have been done on muscle imbalance Lower crossed syndrome (LCS) using Stretching and Muscle energy Technique (MET). Both have shown superior effects when compared to other treatment modalities/techniques. However there is paucity of literature on effectiveness of stretching and MET in management of LCS.

ELIGIBILITY:
Inclusion Criteria:

* LCS pattern in standing position
* Patients having Chronic low back pain
* Age : 20-50 years
* Both male and females
* Positive Prone Hip Extension movement pattern test

Exclusion Criteria:

* Fracture (wedge compression #)
* Inflammatory disorder
* Acute disc bulge
* Lumber instability
* Idiopathic scoliosis
* Patient with Rheumatoid arthritis (RA) and other systemic diseases

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4th week
  It was calculated through Numeric pain rating scale (NPRS) in which 0 was the lowest value with no pain label and 10 was the highest value with worst possible pain label. The Subjects with respect to their pain intensity were asked to mark a level of NPRS.
ROM assessment of iliopsoas | 4th week
  Range of motion (ROM) was taken via goniometer for iliopsoas was measured with double inclinometer.
ROM assessment of rectus femoris | 4th week
  Range of motion (ROM) was taken via goniometer for rectus femoris was measured with double inclinometer.
ROM assessment of hamstrings | 4th week
  Range of motion (ROM) was taken via goniometer for hamstrings was measured with double inclinometer.
ROM assessment of erector spinae | 4th week
  Range of motion (ROM) was taken via goniometer for erector spinae was measured with double inclinometer.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Bibi Zahida Memorial Teaching Hospital NCS, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frank C, Page P, Lardner R. Assessment and treatment of muscle imbalance: the Janda approach: Human kinetics; 2009.
- [Background] Key J, Clift A, Condie F, Harley C. A model of movement dysfunction provides a classification system guiding diagnosis and therapeutic care in spinal pain and related musculoskeletal syndromes: a paradigm shift-Part 1. J Bodyw Mov Ther. 2008 Jan;12(1):7-21. doi: 10.1016/j.jbmt.2007.04.005. Epub 2007 Jun 11. PMID 19083651
- [Background] Kolar P. Facilitation of agonist-antagonist co-activation by reflex stimulation methods. Rehabilitation of the Spine. 2007:531-65.
- [Background] Norkin CC, White DJ. Measurement of joint motion: a guide to goniometry, 5th edition: FA Davis; 2016.
- [Background] Kage MV. Effectiveness of Stretching and Strengthening Exercises in Patients with postural Low Back Pain A Randomized Controlled Trial. 2017.
- [Background] Abutaleb EE, Eldesoky MT, El Rasol SA. Effect of Muscle Energy Technique on Anterior Pelvic Tilt in Lumbar Spondylosis Patients. World Academy of Science, Engineering and Technology, International Journal of Medical, Health, Biomedical, Bioengineering and Pharmaceutical Engineering. 2015;9(8):651-5.
- [Background] Ahmed ET, Abdelkarim SS. Efficacy of muscle energy technique versus static stretching technique in increasing hamstring flexibility post burn contracture. Int J Health Rehabil Sci. 2013;2(1):22-7.